CLINICAL TRIAL: NCT01577277
Title: OPUS(Optimal Well-being, Development and Health for Danish Children Through a Healthy New Nordic Diet) School Meal Study - - Cross Sectional Analyses From Baseline Investigations
Brief Title: OPUS School Meal Study - Cross Sectional Analyses From Baseline Investigations
Status: Completed | Type: Observational
Sponsor: Arne Astrup (Other)
Collaborators: Technical University of Denmark (Other); University of Aarhus (Other); University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Arne Astrup, Professor, MD, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: D208 baseline; H-1-2010-124 (Other: The Regional Committee on Biomedical Research Ethics)
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Metabolic Syndrome X
Keywords: Metabolic Syndrome X; Fatty Acids, Omega-3; Learning; Attention; Nutritional Status; Nutrition Assessments; Body Weight; Physical Activity; Sleep; Child Nutrition Sciences
MeSH Terms: conditions — Metabolic Syndrome; Body Weight; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum and white cells
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study is based on cross-sectional data from the baseline investigations carried out in OPUS School Meal Study - a randomized crossover study carried out in 9 primary schools in Denmark 2011-2012. Approximately 800 Danish school children from 3rd and 4th grades (8-12 year olds) took part in these baseline investigations of socioeconomic status, pubertal status, growth status, learning abilities, well-being, sleep, physical activity and risk markers of Cardiovascular Disease (CVD), type II diabetes and osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Pupils in 3rd and 4th grades
* Primary Schools in the Zealand Region and Capital Region of Denmark Schools with an available school kitchen, that can be approved by the food authorities
* Schools where at least 60 % of the pupils in three or more classes signs up to participate in the Study

Exclusion Criteria:

* The children should not participate in a scientific study or have participated in a scientific study within the last 4 weeks. This, however depends on the character of the other study.
* The children must not suffer from serious food allergies or food intolerance.
* The children must not suffer from diseases or conditions that makes them ill-suited for participation in the study, eg. malabsorptive conditions or serious mental disorders
* The schools must not offer an well-established common meal plan, that provides most of the pupils with healthy food on a daily basis

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: School children participating in OPUS School Meal Study (registered as an intervention study with protocol number: NCT01457794)
Sampling Method: Non-Probability Sample
Enrollment: 834 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome score | Baseline (Cross-sectional)
  The metabolic syndrome score is a continuous z-score based on individual z-scores for Waist Circumference (WC), Mean Arterial Pressure (MAP), serum High Density Lipoprotein (HDL), serum Triglyceride (TG) and Homeostasis Model Assessment (HOMA) index. It´s an internal score meaning that the basis for the score is the distribution of values in this study population.
Body composition | Baseline (Cross-sectional)
  Body composition will be determined by Dual energy X-ray Absorptiometry (DXA) scanning. The parameters included are total body Fat Free Mass Index (FFMI in kg/m2), total body Fat Mass Index (FMI in kg/m2), total body fat percentage and the ratio between android and gynoid fat mass in kg.
Concentration Performance | Baseline (Cross-sectional)
  Concentration Performance is assessed by means of a concentration test called the D2-test of Attention. Concentration Performance is derived from the number of correctly crossed out relevant items minus the errors of commission (confused).
Fatty acid composition in whole-blood | Baseline (cross-sectional)
  Content of saturated fatty acids, monounsaturated fatty acids, polyunsaturated fatty acids, total n-3 and n-6 polyunsaturated fatty acids, eicosapentaenoic acid, docosahexaenoic acid, and the n-6:n-3 ratio in whole-blood measured as weight% relative to the weight of total fatty acids.

SECONDARY OUTCOMES:
Body weight, Body Mass Index (BMI) | Baseline (Cross-sectional)
  Body weight (in kg),BMI, BMI z-score calculated on the basis of the current references from WHO and body weight status (underweight/normal weight/overweight and obese) based on the age and gender specific iso BMI´s defined by Cole et al.
  Cole et al. (2000) BMJ 320 (7244): 1240-1243. Cole et al. (2007) BMJ 335 (7612): 194-197.
Physical activity | Baseline (Cross-sectional)
  Physical activity is measured using waist-worn ActiGraph GT3X and GT3X+. Outcome measures will be counts/min, time spent in sedentary, light, moderate and vigorous activities. The participant are asked to note down non-wear periods in a logbook - mainly to increase compliance - and to note the amount of bicycling and if the child was sick within the measurement period. Questions regarding TV-watching, playing with videogames and physical activity, will help identify activity-pattern.
Sleep | Baseline (Cross-sectional)
  Sleep is measured using ActiGraph GT3X and GT3X+ with the monitor placed on the right hip for all students and on the non-dominant wrist for a sub-sample. Using a sleep diary, total sleep time and sleep quality will be derived from these actigraphy measurements. In addition, the abbreviated version of the Children's Sleep Habits Questionnaire (CSHQ) is used to identify sleep problems.
Cardio-respiratory fitness | Baseline (Cross-sectional)
  Cardio-respiratory fitness is measured using the Andersen test, which is a 10-min intermittent running test to estimate maximal oxygen uptake (mL*min-1*kg-1).
Dietary intake | Baseline (Cross-sectional)
  Dietary intake is measured as micro-and macronutrients as well as food groups (e.g. fish and fruit/vegetables) by means of a 7-day dietary survey, which is a web based recall record method developed especially for children. Families without internet access can use a paper version of a 7-day dietary survey. The meal time perception is measured as well.
Appetite-regulating hormones | Baseline (cross-sectional)
  Leptin and ghrelin. If resources are available at the end of the study period, ghrelin will be separated in acylated and deacylated ghrelin, and both the effect of the intervention on total, acylated, deacylated and the ratio between acylated:deacylated ghrelin will be assessed. If the resources are too tight at the end of the study, only total ghrelin will be used.
Vitamin D status | Baseline (Cross-sectional)
  Serum concentrations of 25-hydroxyvitamin D [25(OH)D] will be used as marker of vitamin D status, related to food intake and time of season.
Bone Health | Baseline (Cross-sectional)
  Bone Health will be evaluated by DXA scanning (total body and spine Bone Mineral Content (BMC), Bone Mineral Density (BMD), and Bone Area (BA). Osteocalcin and serum Parathyreoideahormon (PTH) are also included as markers of bone health.
Iron status | Baseline (Cross-sectional)
  Whole-blood hemoglobin and serum ferritin will be used as measures of iron status
Attention - other measures | Baseline (Cross-sectional)
  The following five measures from the attention test D2 will be used:
  TN=Total Number of items processed E%=Percentage of errors
Wellness | Baseline (Cross-sectional)
  Student wellness is assessed by means of the Danish WRS Wellness Rating Scale filled out by students. The scale contains five subscales and one combined scale (sum score) adding the five subscales. The subscales cover: Living environment, school, school mates, family, and self concept.
Learning | Baseline (Cross-sectional)
  Student learning is assessed by means of the Danish LRS Learning Rating Scale filled out by students. The scale contains four subscales and one combined scale (sum score) adding the four subscales. The subscales cover: Academic learning, social situation in school, teaching style appropriateness, and school expectations.
Mathematics proficiency | Baseline (Cross-sectional)
  Mathematics proficiency is assessed by means of the Danish MG test for 3rd And 4th grade. They each have one measure: Number of correct results within 45 minutes.
Reading proficiency | Baseline (Cross-sectional)
  Reading proficiency is assessed by means of the Danish Sentence Reading test 2 having two measures: Percentage of correct sentences read within eight minutes. Reading speed - number of sentences reached.
Use of ADHD medicine | Baseline (Cross-sectional)
  Among those children with a diagnosis of Attention Deficit/Hyperactivity Disorder (ADHD) or Attention Deficit Disorder (ADD), the mean daily dose of methylphenidate (based on reported intake of drugs containing this substance) during the last two weeks will be evaluated.
Illnesses and use of medicine | Baseline (Cross-sectional)
  Self-reported data collected by personal computer-assisted questionnaire interview with the parents. Outcomes are the number of days, during the last two weeks, with: asthma symptoms, use of asthma-medicine, hay-fever symptoms, use of hay-fever-medicine, atopic eczema, symptoms such as sore throat or fever, and the use of pain killers or antibiotics. The number of days of absence from school due to illness, the number of days of illness during weekends and holidays, and number of visits to the doctor will also be evaluated.
Inflammatory markers | Baseline (Cross-sectional)
  Plasma concentrations of the cytokines Interleucin 6 (IL-6) and Tumor Necrosis factor (TNF-alfa), the adipokine adiponectin and the acute-phase protein C-reative Proetin (CRP)(measured as high-sensitive) in plasma will be used as markers of subclinical inflammation and related to the other early metabolic syndrome and cardiovascular risk markers.
Socioeconomic measures | Baseline (Cross-sectional)
  Self-reported data collected by personal computer-assisted questionnaire interview with the parents. Data are computed on household level. For education and occupation household level = level for the parent or cohabiting partner with the highest value. Education is computed as years of education and as education type. The occupation categorisation is based on the system SOCIO used by Statistics Denmark.
Early Cardiovascular Risk Markers | Baseline (Cross-sectional)
  Systolic and diastolic blood pressure, serum blood cholesterol (total, LDL, VLDL and HDL) and triglyceride, plasma glucose, serum insulin and the HOMA index.
Pubertal status | cross-sectional (baseline)
  Pubertal status is assessed by menstruation status (menstruation started or not) and breast development in girls (Tanner stage 1-5) and by development of pubic hair in boys (Tanner stage 1-5).

OTHER OUTCOMES:
Genotyping | Baseline (Cross-sectional)
  SNPs in genes related to metabolic pathways, messenger molecules, receptors or other genes that may affect efficacy measures in OPUS School Food Project

CONTACTS AND LOCATIONS:
Overall Officials: Kim F Michaelsen, Professor MD, Principal Investigator — Department of Human Nutrition, Faculty of Science, University of Copenhagen Copenhagen, Denmark
Locations (1):
- Department of Human Nutrition, Faculty of Life Sciences, University of Copenhagen Copenhagen, Denmark, Copenhagen, Denmark

REFERENCES:
- [Derived] Damsgaard CT, Biltoft-Jensen A, Tetens I, Michaelsen KF, Lind MV, Astrup A, Landberg R. Whole-Grain Intake, Reflected by Dietary Records and Biomarkers, Is Inversely Associated with Circulating Insulin and Other Cardiometabolic Markers in 8- to 11-Year-Old Children. J Nutr. 2017 May;147(5):816-824. doi: 10.3945/jn.116.244624. Epub 2017 Mar 29. PMID 28356426